CLINICAL TRIAL: NCT00002738
Title: Phase II Trial of Trimetrexate and Leucovorin in The Treatment of Recurrent Childhood Acute Lymphoblastic Leukemia
Brief Title: Combination Chemotherapy in Treating Children With Acute Lymphoblastic Leukemia, Osteosarcoma, or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 95-093; P30CA008748 (NIH); MSKCC-95093; NCI-V96-0840
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Leukemia; Lymphoma; Sarcoma
Keywords: recurrent childhood acute lymphoblastic leukemia; recurrent childhood lymphoblastic lymphoma; recurrent osteosarcoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Sarcoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Osteosarcoma; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating | interventions — Leucovorin; trimetrexate glucuronate

INTERVENTIONS:
Drug: leucovorin calcium
Drug: trimetrexate glucuronate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as trimetrexate glucuronate and leucovorin, use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: This phase II trial is studying how well combination chemotherapy works in treating children with recurrent acute lymphoblastic leukemia, recurrent osteosarcoma, or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of trimetrexate glucuronate with leucovorin calcium rescue in children with recurrent acute lymphoblastic leukemia, recurrent osteogenic sarcoma, or refractory non-Hodgkin's lymphoma resistant to methotrexate.
* Evaluate the toxicity of this treatment regimen in this patient population.

OUTLINE: Patients are stratified according to disease (acute lymphocytic leukemia, non-Hodgkin's lymphoma vs osteogenic sarcoma).

Patients receive trimetrexate glucuronate orally or IV every 12 hours on days 1-21 and oral leucovorin calcium every 12 hours on days 1-24. Treatment repeats every 4 weeks. Patients with stable or responsive disease may receive up to 4 courses of therapy.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologic evidence of one of the following malignancies that has failed conventional therapy:

  * Acute lymphoblastic leukemia
  * Non-Hodgkin's lymphoma with bone marrow involvement
  * Osteogenic sarcoma
* In vitro transport resistance to methotrexate demonstrated by bone marrow aspirate assay

PATIENT CHARACTERISTICS:

Age:

* 21 and under at diagnosis

Performance status:

* ECOG 0-2

Life expectancy:

* At least 8 weeks

Hematopoietic:

* Granulocytopenia allowed with bone marrow involvement
* Thrombocytopenia allowed with bone marrow involvement
* Anemia allowed with bone marrow involvement

Hepatic:

* (unless due to disease)
* Bilirubin no greater than 2.0 mg/dL
* AST no greater than 100

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Other:

* No other serious medical illness
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior bone marrow transplantation allowed

Chemotherapy:

* At least 1 week since prior intrathecal treatment
* At least 2 weeks since prior systemic chemotherapy and recovered

  * At least 10 days for rapidly proliferating leukemia (i.e., WBC greater than 50,000)
* No concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior radiotherapy allowed and recovered
* No concurrent radiotherapy

Surgery:

* Not specified

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 1996-01; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Trippett, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States